CLINICAL TRIAL: NCT05127382
Title: Osimertinib as First Line Therapy for Patients With Advanced EGFR Positive Non-Small Cell Lung Cancer: the Experience of the Hellenic Cooperative Oncology Group (HeCOG)
Brief Title: Osimertinib as 1st Line Therapy for Patients With Advanced EGFR Positive Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE219
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer Non-small Cell Stage IV
Keywords: non-small cell lung cancer; egfr mutation; osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be collected from patients with advanced egfr positive non-small cell lung cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- untreated patients with advanced EGFR positive non-small cell lung cancer

SUMMARY:
The present study will evaluate the use of osimertinib as 1st line therapy for patients with advanced EGFR positive non-small cell lung cancer who are treated at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology.

DETAILED DESCRIPTION:
This will be an observational, multicentric, retrospective/ prospective analysis of patients with advanced EGFR positive non-small cell lung cancer that receive osimertinib as 1st line therapy. The patient data will be collected at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology during scheduled patient clinical visits, from February 2020 for a total period of three years. The biological material obtained from the patients of this analysis will be possibly used in a future translational study as an exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* men or women of 18 years or older that live in Greece
* histologically or cytologically confirmed, advanced EGFR positive non-small cell lung cancer
* untreated patients for advanced NSCLC
* patients who are expected to receive osimertinib regardless of their enrollment in the study
* signed written informed consent

Exclusion Criteria:

* patients with cancer other than NSCLC that require treatment
* pretreated patients for NSCLC
* patients that receive or are expected to receive or have received an investigational drug/product/intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced EGFR positive non-small cell lung cancer that receive osimertinib as 1st line therapy and are treated at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | through the completion of the study, up to 2 years
  the time from treatment initiation to either the first documented disease progression or death from any cause

SECONDARY OUTCOMES:
overall survival (OS) | through the completion of the study, up to 2 years
  the time from treatment initiation to patient death or last contact
overall response rate (ORR) | through the completion of the study, up to 2 years
  the response rate for all enrolled population and for the response evaluable population
quality of life data | through the completion of the study, up to 2 years
  quality of life data through EQ-5D-5L questionnaire
Safety profile and toxicity | through the completion of the study, up to 2 years
  Rates of adverse events because of treatment with osimertinib
health economics | through the completion of the study, up to 2 years
  description of health costs to determine cost-effectiveness of osimertinib
second progression-free survival (PFS2) | through the completion of the study, up to 2 years
  time from treatment initiation to objective tumour progression on next-line treatment or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Cooperative Oncology Group, Athens, Greece